CLINICAL TRIAL: NCT04902456
Title: Evaluation of the Anchorage Loss During En-masse Retraction in Orthodontic Patients With Maxillary Protrusion Using Friction Versus Frictionless Mechanics: A Randomized Clinical Trial
Brief Title: Evaluation of the Anchorage Loss During En-masse Retraction in Orthodontic Patients With Maxillary Protrusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Amr Mahmoud Attia, Principle Investigator, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUE.REC (13)/7-2019
Record Dates: First submitted 2021-05-15; First posted 2021-05-26 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Bimaxillary Protrusion
Keywords: En-masse Retraction; Friction; Frictionless; CBCT; Anchorage; Anchorage loss; Dental models

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Only the outcome assessors will be blind. The patients name will be sealed from pre and post radiographs and study models. Then two assessors will carry out, blindly and independently, the measurements and analysis of the study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Power Chain and Crimpable hook for En-masse retraction (Experimental): Retraction will start on a 0.017x0.025" Stainless Steel wire using elastomeric chain ( force applied will be 212 g per side ) extending between the crimpable hooks and the miniscrew
  Interventions: Procedure: Power chain and Crimpable hook fro En-masse Retraction
- T-loop (Experimental): Closing retraction T-loops will be fabricated using 0.017x0.025" TMA wire. The loop will be positioned halfway the extraction space and the canine.
  Interventions: Procedure: T-loop

INTERVENTIONS:
Procedure: Power chain and Crimpable hook fro En-masse Retraction — Retraction will start on a 0.017x0.025" stainless steel wire using elastomeric chain ( for applied will be 212 g per side ) extending between the cripmable hooks and the miniscrew
  Arms: Power Chain and Crimpable hook for En-masse retraction
Procedure: T-loop — closing retraction T-loops will be fabricated using 0.017x0.025 TMA wire. The loop will be positioned halfway the extraction space and the canine.
  Arms: T-loop

SUMMARY:
There is scarcity in literature regarding the effectiveness of friction and frictionless mechanics during ''En-masse retraction''technique on anchorage loss of posterior segment in orthodontic patients with maxillary protrusion. Moreover there is deficiency in studies measuring the patient pain and satisfaction regarding the different techniques of retraction.

The aim of the current study is to evaluate the effects of friction versus frictionless mechanics, implemented during "En-masse retraction", on anchorage loss. Additionally, assessment of both techniques regarding their rates, effects on root resorption as well as patient satisfaction.

DETAILED DESCRIPTION:
One of the most common complaints of orthodontic patients is proclination of anterior teeth where there is an increase in facial convexity and as well as incompetent lips. Bimaxillary dentoalveolar protrusion and class II division I cases always have this appearance. Frequently this situation requires extraction of the first premolars followed by fixed orthodontic appliance for space closure and retraction of anterior teeth. Different techniques are used including "Two-step retraction" where canines are retracted as a first step followed by anterior four incisors as a second step and "En-masse retraction" where anterior teeth are retracted as one unit. However, the method of "En-masse retraction" is controversial - whether to use frictionless or friction mechanics.

ELIGIBILITY:
Inclusion Criteria:

1. Orthodontic patients (both genders)
2. Age range (14-24)
3. Patients requiring 1st premolars extraction followed by ''En-masse retraction'' (Bimaxillary Protrusion or Class II division 1 cases).
4. Patients with fully erupted permanent teeth (not necessarily including the 3rd molar).
5. Cases requiring maximum anchorage during anterior segment retraction.
6. Cases with minimal crowding (2-3) mm

Exclusion Criteria:

1. Patients suffering from any systemic diseases interfering with tooth movement.
2. Patients with extracted or missing permanent teeth. (except for third molars).
3. Patients with badly decayed teeth.
4. Patients with any parafunctional habits (i.e. Bruxism, tongue thrusting, mouth breathing, etc....).
5. Patients with previous orthodontic treatment

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2022-01-29 (Estimated); Study Completion 2022-01-29 (Estimated)

PRIMARY OUTCOMES:
Anchorage loss | from pre to post retraction/intervention ( an average of 6-8 months )
  Digitally scanned dental models taken pre and post completion of retraction will be measured by identifying landmarks and reference lines and planes ( measured in mm )

SECONDARY OUTCOMES:
Retraction Rate | from pre to post retraction/intervention ( an average of 6-8 months )
  The antero-posterior movement of anterior teeth and first molars will be assessed by measuring the digitally scanned dental models taken of the patients monthly ( measured in mm )
Molar Rotation | from pre to post retraction/intervention ( an average of 6-8 months )
  Digitally scanned dental models that are taken before and after retraction will be assess the rotation of the maxillary first permanent molar in relation to a reference line ( measurement of the angles in degrees )
Pain of Intervention | from pre to post retraction/intervention ( an average of 6-8 months )
  each patient will fill a questionnaire regarding his treatment experience in a Visual Analog Scale (VAS) scoring from 1-10 by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10 cm). The question-naire will include several questions related to oral hygiene, pain and discomfort experienced throughout the trial.
Anterior teeth extrusion/intrusion | from pre to post retraction/intervention ( an average of 6-8 months )
  The principle investigator will examine pre and post Cone Beam CT ( CBCT ) in Relation to lines and reference planes ( measured in mm )
Anterior teeth torque | from pre to post retraction/intervention ( an average of 6-8 months )
  The principle investigator will examine pre and post Cone Beam CT ( CBCT ) in Relation to lines and reference planes ( measured in degrees )
Anterior teeth tip | from pre to post retraction/intervention ( an average of 6-8 months )
  The principle investigator will examine pre and post Cone Beam CT ( CBCT ) in Relation to lines and reference planes ( measured in degrees )

CONTACTS AND LOCATIONS:
Overall Officials: Yehia Mostafa, Professor and Chairman, Study Director — Future University in Egypt
Locations (1):
- Amr Attia, Cairo, Future University in Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after Publication

DOCUMENTS (2):
  • Study Protocol (2019-12-31): https://cdn.clinicaltrials.gov/large-docs/56/NCT04902456/Prot_000.pdf
  • Informed Consent Form (2019-12-31): https://cdn.clinicaltrials.gov/large-docs/56/NCT04902456/ICF_001.pdf